CLINICAL TRIAL: NCT06645899
Title: Creation, Management and Analysis of a National Database of Patients Affected by Hypoparathyroidism or Pseudohypoparathyroidism
Brief Title: Institution of an Italian Multicenter Database of Patients Affected by Hypoparathyroidism or Pseudohypoparathyroidism
Status: Recruiting | Type: Observational
Sponsor: F.I.R.M.O. - Fondazione Italiana Ricerca sulle Malattie dell'Osso - Ente del Terzo Settore (Other)
Responsible Party: Sponsor
Other Study IDs: 23235_oss
Record Dates: First submitted 2024-10-07; First posted 2024-10-17 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2024-10

CONDITIONS: Hypoparathyroidism; Pseudo Hypoparathyroidism
Keywords: Hypoparathyroidism; Pseudohypoparathyroidism; Database of patients; Retro-prospective clinical data collection
MeSH Terms: conditions — Hypoparathyroidism; Pseudohypoparathyroidism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with hypoparathyroidism: Male and female patients of any age who are affected by chronic hypoparathyroidism.
  The observation study does not include any type of intervention.
- Patients with pseudohypoparathyroidism: Male and female patients of any age who are affected by pseudohypoparathyroidism.
  The observation study does not include any type of intervention.

SUMMARY:
The goal of this observational study is to create, manage and analyze a multicenter national database of patients affected by hypoparathyroidism or pseudohypoparathyroidism, aimed at collecting and studying anamnestic, diagnostic, genetic, clinical, and therapeutic data in a relatively wide number of patients with these two rare pathologies, in Italy.

The study will include 41 specialist clinical centers of endocrinology, pediatric endocrinology, pediatrics, and endocrine surgery, located throughout the Italian territory, and to which patients refer from all the 20 regions of Italy.

Data will be collected over time, both in retrospective and prospective manners, during the 10-year duration of the study, starting from the recruiting visit (basal visit) and then during each follow-up visits patients will undergo for the control of disease at the recruiting clinical centers.

Collected data will include both the most classic traits of the pathology and the less common ones, with the final goal of refining and deepening medical knowledge in the field of these two clinical conditions affecting parathyroid function and calcium homeostasis, and, thus, to be able to define optimal clinical and therapeutic management of patients, improving their quality of life.

The main aspects this observational study aims to assess and clarify are:

1. Evaluation of prevalence and incidence of hypoparathyroidism, globally and in its different etiological forms, and of pseudohypoparathyroidism in Italy.
2. Clinical characterization of different etiological forms of hypoparathyroidism, through both cross-sectional and longitudinal analyses of collected data.
3. Clinical characterization of pseudohypoparathyroidism, through both cross-sectional and longitudinal analyses of collected data.
4. Over time collection of data on bone status and bone fragility in patients with hypoparathyroidism and pseudohypoparathyroidism, to evaluate the prevalence and incidence of fragility fractures in these patients, globally and also based on gender, age, and disease etiology.
5. Over time evaluation of response to pharmacological therapies in patients with hypoparathyroidism and pseudohypoparathyroidism The study will include two independent cohorts of female and male patients of any age, one including patients with chronic hypoparathyroidism of each etiological forms (cohort 1), and one including patients with pseudohypoparathyroidism (cohort 2). The study does not include either any control group/comparison group or healthy volunteers.

The study itself does not involve any medical intervention or drug administration. Pharmacological treatments for which data on response to therapy will be collected in the database, are those administered to patients for the control/treatment of hypoparathyroidism or pseudohypoparathyroidism, regardless of their inclusion in this observational study.

DETAILED DESCRIPTION:
A. Background and rationale:

Hypoparathyroidism is a rare endocrine disease characterized by low levels of calcium (hypocalcemia) and high levels of phosphorus (hyperphosphatemia) in the blood, as a result of inappropriately low or completely absent levels of parathyroid hormone (PTH). Data on the global epidemiology of this disease are still incomplete, it is estimated to affect less than 1 case in 200,000 people. Even more incomplete are the national incidence data.

Hypoparathyroidism can be acquired or congenital. The most common form of hypoparathyroidism is post-surgical (about 75% of cases), following surgery in the neck region with damage and/or removal of the parathyroid glands. Among other forms of acquired hypoparathyroidism there are, in a much lower percentage, those caused by irradiation of the neck, viral infections with infiltration of the parathyroid tissue (i.e. tuberculosis), metastatic infiltrations, autoimmune diseases, chronic magnesium depletion (malabsorption, alcoholism or malnutrition).

Congenital hypoparathyroidism can be caused by germline mutations in various genes, which regulate the correct development and/or functionality of the parathyroid glands and synthesis and release of PTH, and can arise as an isolated or syndromic form, the latter in association with other endocrine and non-endocrine alterations.

The term pseudohypoparathyroidism, on the other hand, refers to a heterogeneous group of hereditary diseases characterized by resistance to PTH in target organs (proximal tubules of the kidney), which causes hypocalcemia and hyperphosphatemia in the presence of normal and even elevated PTH levels.

The real global and Italian prevalence and incidence of hypoparathyroidism and pseudohypoparathyroidism is not certain; the lack of specific national and international registries for this pathology remains a major limitation to its in-depth clinical understanding and to the optimization of the therapeutic management of patients.

Implementing and detailing as much as possible the epidemiological, clinical and therapeutic history of hypoparathyroidism, in its various etiological forms, and pseudohypoparathyroidism means not only improving the clinical management of the individual patient, but also allowing for better planning of social, political and health interventions for these pathologies and, overall, improving the quality and life expectancy of patients.

For this reason, it is extremely important to create multicenter national databases, such as the one proposed by this study, which allow to collect a relatively high number of patients affected by hypoparathyroidism or pseudohypoparathyroidism, whose cases can be, thus, carefully studied in every aspect, both retrospectively and prospectively.

A previous Italian database (HypoparaNET) [1] was established in the period March 2014-September 2015, collecting 509 cases of chronic hypoparathyroidism from 16 Italian Endocrinological Clinical Centers. However, this database collected patients' data limited exclusively to the time of inclusion in the study, not including the collection of follow-up data, and, thus, allowing only an epidemiological evaluation and a cross-sectional observational analysis of the data collected at the time of inclusion in the study.

Instead, in the present study, the investigators aim to collect data on hypoparathyroidism and pseudohypoparathyroidism cases over time, allowing not only to analyze epidemiological data and to perform a single shot analysis of collected data, but also to be able to perform longitudinal analyses of the two diseases, with particular attention to the response to therapies.

B. Main aim and specific objectives:

Main goal of this observational study is to create, manage and analyze a retro-prospective multicenter national database of patients with hypoparathyroidism or pseudohypoparathyroidism in Italy, aimed at collecting and studying anamnestic, diagnostic, genetic, clinical, and therapeutic data on these two endocrine diseases in a relatively wide number of patients.

Such a database will allow for an epidemiological evaluation of prevalence and incidence hypoparathyroidism or pseudohypoparathyroidism in Italy, and to collect case history of patients whose clinical cases will be studied in detail and followed over time up to 10 years after the recruitment in the study, in order to refine knowledge in the field of these two rare endocrine diseases.

Specific objectives of the studies are:

1. Creation of an Italian centralized multicenter database of patients with hypoparathyroidism or pseudohypoparathyroidism, through the collection of patients at 41 specialist clinical centers of endocrinology, pediatric endocrinology, pediatrics, and endocrine surgery, located throughout the Italian territory and visiting patients from all the 20 regions of Italy.
2. Collection of a relatively high number of patients with hypoparathyroidism of different etiology or with pseudohypoparathyroidism.
3. Retrospective collection of data about hypoparathyroidism or pseudohypoparathyroidism, at the time of the recruiting visit.
4. Continuous and updated prospective collection of patients' data over time, starting from the first recruiting visit up to 10 years after the recruitment in the study.
5. Evaluation of prevalence and incidence of hypoparathyroidism, globally and in its different etiological forms, and of pseudohypoparathyroidism, in Italy.
6. Clinical characterization of different etiological forms of hypoparathyroidism, through both cross-sectional and longitudinal analyses of collected data
7. Clinical characterization of pseudohypoparathyroidism, through both cross-sectional and longitudinal analyses of collected data
8. Over time collection of data on bone status and bone fragility in patients with hypoparathyroidism and pseudohypoparathyroidism, to evaluate the prevalence and incidence of fragility fractures in these patients also based on gender, age, and disease etiology
9. Over time evaluation of response to pharmacological therapies in patients with hypoparathyroidism and pseudohypoparathyroidism.

C. Study population:

The study will include two independent cohorts of female and male patients of any age, one including patients with chronic hypoparathyroidism (cohort 1), and one including patients with pseudohypoparathyroidism (cohort 2).

The study does not include either any control group/comparison group or healthy volunteers.

Based on the previous experience with the HypoparaNET database, the investigators can estimate to be able to include in the study at least 600 patients affected by hypoparathyroidism or pseudohypoparathyroidism during the 10 years of the study.

Inclusion criteria

* Cohort 1: chronic hypoparathyroidism (all etiological forms)
* Cohort 2: pseudohypoparathyroidism Exclusion criteria
* None

D. Study design and setting:

Non-profit, multicenter, national, retro-prospective, observational study, consisting in the design, creation, management and analysis of an Italian database of patients with hypoparathyroidism or pseudohypoparathyroidism.

The study will last 10 years. The enrollment of patients with hypoparathyroidism or pseudohypoparathyroidism, the inclusion in the database with retrospective collection of their clinical data, and the subsequent prospective collection of clinical follow-up data will take place throughout the duration of the study. For the retrospective collection, retrospective data on hypoparathyroidism or pseudohypoparathyroidism will be retrieved from patient's medical records, at the time of the medical visit that the patient will carry out at the Clinical Center for the evaluation of his/her disease, regardless of inclusion in this study. Prospective data relating to hypoparathyroidism or pseudohypoparathyroidism follow-up will be collected during the subsequent medical follow-up visits, scheduled for each patient as part of the clinical management of his/her clinical condition, regardless of inclusion in this study.

Being an observational study, this study itself does not involve the administration of any drug, nor the use of any medical device, nor does it involve additional medical visits, clinical analyses or care procedures in addition to those conventionally scheduled for the clinical and therapeutic management of patient affected by hypoparathyroidism or pseudohypoparathyroidism. No participant biospecimens of any type will be collected and retained to perform this study. Pharmacological treatments for which data on response to therapy will be collected in the database, are those usually administered to patients for the control/treatment of hypoparathyroidism or pseudohypoparathyroidism, regardless of their inclusion in this observational study.

All data will be collected anonymously, and they will be analyzed as aggregates. Data collected in the database will be, first, processed using descriptive statistics, such as frequency tables for categorical data, median and quartiles for quantitative data on ordinal scales and mean and standard deviation for quantitative data on metric scales. Secondly, the correlations between variables will be evaluated using the Pearson correlation index in the case of continuous variables and the chi-square test for categorical variables.

E. Data and variables:

Data collected in the database will include (if available in patient's medical records and part of the normal clinical and therapeutic management of patient regardless of inclusion in this study):

* Demographics (sex, year of birth)
* Family history of chronic hypoparathyroidism or pseudohypoparathyroidism in first-degree relatives (only for patients with a congenital form of the disease)
* History of neck irradiation, viral infections with infiltration of the parathyroid tissue (i.e. tuberculosis), metastatic infiltrations, autoimmune diseases, chronic magnesium depletion, and neck surgery as possible cause of chronic hypoparathyroidism
* Presence of comorbidities
* Age at diagnosis/onset of hypoparathyroidism or pseudohypoparathyroidism
* Genetic testing for congenital forms of hypoparathyroidism or pseudohypoparathyroidism (if performed)
* Clinical manifestations of the diseases (i.e paresthesia, cramps, tetany, chondrocalcinosis, nephrocalcinosis, nephrolithiasis, chronic renal failure, ectopic calcifications, neurocognitive and brain disorders, ocular manifestations)
* DXA and/or pQCT/HR-pQCT evaluation of bone status
* History of fragility fractures
* Biochemical measurements of parameters of parathyroid function, bone and mineral metabolism and renal function (at baseline and follow-up visits)
* Pharmacological therapies (drug, duration, posology)
* Self-evaluation of quality of life (i.e. Questionnaire SF36)
* Disease-related morbidity and mortality

ELIGIBILITY:
Inclusion Criteria:

* Cohort 1: chronic hypoparathyroidism (all etiological forms)
* Cohort 2: pseudohypoparathyroidism

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Two independent cohorts of female and male patients of any age, one including patients with chronic hypoparathyroidism (cohort 1), and one including patients with pseudohypoparathyroidism (cohort 2).
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2034-11-04 (Estimated); Study Completion 2034-11-04 (Estimated)

PRIMARY OUTCOMES:
Prevalence and incidence evaluation | Through study completion, an average of 10 years
  Evaluation of prevalence and incidence of hypoparathyroidism globally and in its different etiological forms, and of pseudohypoparathyroidism in Italy
Clinical characterization of hypoparathyroidism | Through study completion, an average of 10 years
  Clinical characterization of different etiological forms of hypoparathyroidism, through both cross-sectional and longitudinal analyses of collected data
Clinical characterization of pseudohypoparathyroidism | Through study completion, an average of 10 years
  Clinical characterization of pseudohypoparathyroidism, through both cross-sectional and longitudinal analyses of collected data
Bone fragility in patients with hypoparathyroidism and pseudohypoparathyroidism | Through study completion, an average of 10 years
  Evaluation of over time prevalence and incidence of fragility fractures in patients with hypoparathyroidism and pseudohypoparathyroidism, globally and also based on gender, age, and disease etiology
Therapy response in patients with hypoparathyroidism and pseudohypoparathyroidism | Through study completion, an average of 10 years
  Over time analysis of responses to pharmacological therapies in in patients with hypoparathyroidism and pseudohypoparathyroidism

CONTACTS AND LOCATIONS:
Locations (41):
- Italy (41):
  - SC Pediatria e Pronto Soccorso Pediatrico - AOU SS. Antonio e Biagio e C. Arrigo, Alessandria
  - U.O.C. Endocrinologia, Azienda Ospedaliero Universitaria Policlinico Consorziale, Università degli Studi di Bari "Aldo Moro", Bari
  - Unità di Pediatria, IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna
  - UOC Endocrinologia e Prevenzione e Cura del Diabete, IRCCS Azienda Ospedaliero-Universitaria di Bologna, Dipartimento di Scienze Mediche e Chirurgiche (DIMEC), Alma Mater Studiorum Università di Bologna, Bologna
  - Centro di Auxoendocrinologia e Genetica Medica della Clinica Pediatrica degli Spedali Civili di Brescia, Brescia
  - Endocrinologia e Diabetologia, Azienda Ospedaliero-Universitaria di Cagliari, Presidio Ospedaliero Policlinico di Monserrato, Cagliari
  - UO Endocrinologia e Malattie del Ricambio, Azienda Ospedaliero Universitaria di Ferrara, Sezione di Endocrinologia, Geriatria e Medicina Interna, Dipartimento di Scienze Mediche, Università degli Studi di Ferrara, Ferrara
  - Diabetologia e Endocrinologia, Auxoendocrinologia, Children's Hospital Meyer IRCCS, Florence
  - SOD Malattie del Metabolismo Minerale ed Osseo, Azienda Ospedaliero-Universitaria Careggi, Florence
  - Ospedale Casa Sollievo della Sofferenza, Foggia
  - Centro di Alta Specialità in Osteoporosi Pediatrica e Malattie del Metabolismo Calcio-Fosforo, U.O.C. Clinica Pediatrica, Dipartimento di Scienze Pediatriche Generali e Specialistiche IRCCS Istituto Giannina Gaslini, Genova
  - Clinica Endocrinologica, Dipartimento di Medicina Interna e Specialità Mediche (DiMI), IRCCS Ospedale Policlinico San Martino, Università di Genova, Genova
  - U.O.S.D. Centro Malattie Rare · Dipartimento di Pediatria IRCCS Ospedale Pediatrico Giannina Gaslini, Genova
  - Dipartimento di Patologia Umana dell'adulto e dell'età evolutiva "Gaetano Barresi", Università degli Studi di Messina, Messina
  - UOC di Endocrinologia, AOU Policlinico G. Martino, Dipartimento di Patologia Umana DETEV, Università di Messina, Messina
  - Dipartimento di Malattie Endocrino-Metaboliche, IRCCS Istituto Auxologico Italiano, Milan
  - Endocrinologia Infantile, UOU di Pediatria, IRCCS Ospedale San Raffaele, Milan
  - IRCCS Ospedale San Raffaele, Milan
  - SC Endocrinologia, Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Dipartimento di Medicina Clinica e Chirurgia; Unità di Endocrinologia, Diabetologia e Andrologia; Università degli Studi di Napoli Federico II, Napoli
  - UOC di Endocrinologia e Malattie del Metabolismo, AOU Università degli Studi della Campania Luigi Vanvitelli, Napoli
  - UOS di Endocrinologia Pediatrica, Dipartimento Materno Infantile, AOU Federico II, Napoli
  - UOSD Malattie Neuro-Endocrine, Centro Obesità, Dipartimento di Neuroscienze e Riabilitazione, AORN Santobono-Pausilipon, Napoli
  - SCDU Endocrinologia Azienda Ospedaliero-Universitaria Maggiore della Carità di Novara, Novara
  - Endocrinologia, Clinica Polispecialistica San Carlo, Paderno Dugnano
  - Unità di Chirurgia Endocrina, Dipartimento di Chirurgia, Oncologia e Gastroenterologia, Università di Padova, Padua
  - UOC Endocrinologia, DIMED, Azienda Ospedaliero-Universitaria di Padova, Padua
  - Unità Operativa Endocrinologia 2, Azienda Ospedaliera Universitaria Pisana, Pisa
  - Dipartimento di Medicina Sperimentale, "Sapienza" Università di Roma, Roma - UOC Endocrinologia, Policlinico Umberto I di Roma, Roma
  - Unità di Endocrinologia e Andrologia, Dipartimento di Medicina Clinica e Molecolare, AOU Sant'Andrea, Centro di eccellenza ENETS, Università Sapienza di Roma, Roma
  - UOC di Endocrinologia e Diabetologia, UOS di Endocrinologia Pediatrica, IRCCS Ospedale Pediatrico Bambino Gesù, Roma
  - UOC Patologie osteo-metaboliche e della tiroide, Fondazione Policlinico universitario Campus Bio-Medico, Roma
  - UOC di Endocrinologia, Diabetologia e Andrologia Medica, IRCCS Humanitas Research Hospital, Rozzano
  - Donatello Bone Clinic, Casa di Cura Villa Donatello, Sesto Fiorentino
  - Dipartimento di Scienze Mediche, Chirurgiche e Neuroscienze, Policlinico Santa Maria delle Scotte, Università di Siena, Siena
  - Endocrinologia Pediatrica Ospedale Infantile regina Margherita-Dipartimento di Scienze di Sanità Pubblica e Pediatriche, Università degli studi di Torino, Torino
  - SCDU Endocrinologia Diabetologia e Malattie del Metabolismo, AOU Città della Salute e della Scienza di Torino, Università di Torino, Torino
  - SCDU Endocrinologia Oncologica, AOU Città della Salute e della Scienza di Torino, Università di Torino, Torino
  - IRCCS Materno-Infantile Burlo Garofolo, Trieste
  - SOC Endocrinologia, Azienda Sanitaria-Universitaria Friuli Centrale, Udine
  - UOS di Endocrinologia, Policlinico GB Rossi, Azienda Ospedaliera Universitaria Integrata di Verona, Verona